CLINICAL TRIAL: NCT02406586
Title: Free Fatty Acids-Induced Hypertension, Endothelial Dysfunction, Inflammation, Insulin Resistance, and Autonomic Dysfunction in Lean and Obese Subjects (Aim #2)
Brief Title: Free Fatty Acids-Induced Hypertension in Obese Subjects (Aim #2)
Acronym: FFAADA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, MD, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00009277a
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Results first posted 2015-05-28 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Hypertension; Diabetes
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — salicylsalicylic acid; Anti-Inflammatory Agents, Non-Steroidal; Carvedilol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Salsalate (Experimental): Obese, normotensive, healthy subjects will receive an intravenous (IV) administration of Intralipid 20% for 24 hours, and then one salsalate 750 mg tablet twice daily for two weeks. If the subject has no side effects, the dose will be increased to two salsalate 750 mg tablets twice daily for the remaining four weeks. The subjects will then receive another 24-hour IV administration of Intralipid 20% at the 6-week point.
  Interventions: Drug: Salsalate; Drug: Intralipid 20%
- Carvedilol (Experimental): Obese, normotensive, healthy subjects will receive an intravenous (IV) administration of Intralipid 20% for 24 hours, and then one carvedilol 3.125 mg tablet twice daily for two weeks. If the subject has no side effects, the dose will be increased to two carvedilol 3.125 mg tablets twice daily for the remaining four weeks. The subjects will then receive another 24-hour IV administration of Intralipid 20% at the 6-week point.
  Interventions: Drug: Carvedilol; Drug: Intralipid 20%
- Placebo (Placebo Comparator): Obese, normotensive, healthy subjects will receive an intravenous (IV) administration of Intralipid 20% for 24 hours, and then one placebo tablet twice daily for two weeks. The dose will be increased to two placebo tablets twice daily for the remaining four weeks. The subjects will then receive another 24-hour IV administration of Intralipid 20% at the 6-week point.
  Interventions: Drug: Placebo; Drug: Intralipid 20%

INTERVENTIONS:
Drug: Salsalate — Salsalate 750 mg
  Other Names: Disalcid; NSAID
  Arms: Salsalate
Drug: Carvedilol — Carvedilol 3.125 mg
  Other Names: Coreg
  Arms: Carvedilol
Drug: Placebo — One tablet
  Arms: Placebo
Drug: Intralipid 20% — 24-hour infusion of Intralipid 20% solution at 20 mL/h (96 g/24 h)
  Other Names: 20% I.V. Fat Emulsion

SUMMARY:
The purpose of this study is to see if salsalate, an Nuclear factor-kappaB (NF-κB) mediated inflammation inhibitor, or carvedilol, an α- and β-blocker, will protect against free fatty acid induced hypertension, insulin resistance, endothelial dysfunction, inflammation and oxidative stress, and autonomic dysfunction in obese normotensive subjects.

DETAILED DESCRIPTION:
During postprandial lipemia, dietary triglycerides transported by intestinal chylomicrons are hydrolyzed by lipoprotein lipase lining the vascular bed, with subsequent release of FFA for transport across the endothelium. Whether the intermittent flux of FFA has the same impact as the i.v. lipid infusion will be examined. Decreased endothelial function has been reported after a single or long-term dietary high fat load in normal subjects; however, others have found no effects on brachial artery vasoreactivity. Our preliminary studies indicate that high oral fat loads (60 g) resulted in higher FFA levels and BP changes, and reduced FMD compared to low fat load (25 g).

ELIGIBILITY:
Inclusion Criteria:

* Males or females
* Obese subjects (body mass index (BMI) ≥ 30 kg/m^2)
* 18 and 65 years
* Blood pressure reading < 140/80 mm Hg and no prior history of hypertension

Exclusion Criteria:

* History of diabetes mellitus
* History of hypertension
* Fasting triglyceride levels > 250 mg/dL
* Liver disease (ALT 2.5x > upper limit of normal)
* Serum creatinine ≥1.5 mg/dL
* Smokers, drug or alcohol abuse
* Mental condition rendering the subject unable to understand the scope and possible consequences of the study
* Female subjects who are pregnant or breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from July 2009 to January 2011 at Grady Memorial Hospital.
Pre-assignment Details: All subjects will receive IV Intralipid (20% solution at 20 ml/hour) prior to randomization.
Groups:
- Salsalate: Obese, normotensive, healthy subjects received an intravenous (IV) administration of Intralipid 20% for 24 hours, and then one salsalate 750 mg tablet twice daily for two weeks. If the subject had no side effects, the dose was increased to two salsalate 750 mg tablets twice daily for the remaining four weeks. The subjects also received another 24-hour IV administration of Intralipid 20% at the 6-week point.
- Carvedilol: Obese, normotensive, healthy subjects received an intravenous (IV) administration of Intralipid 20% for 24 hours, and then one carvedilol 3.125 mg tablet twice daily for two weeks. If the subject had no side effects, the dose was increased to two carvedilol 3.125 mg tablets twice daily for the remaining four weeks. The subjects also received another 24-hour IV administration of Intralipid 20% at the 6-week point.
- Placebo: Obese, normotensive, healthy subjects received an intravenous (IV) administration of Intralipid 20% for 24 hours, and then one placebo tablet twice daily for two weeks. The dose was increased to two placebo tablets twice daily for the remaining four weeks. The subjects also receive another 24-hour IV administration of Intralipid 20% at the 6-week point.
Period: Overall Study
Arm/Group | Salsalate | Carvedilol | Placebo
Started | 12 | 12 | 12
Completed | 11 | 8 | 10
Not Completed | 1 | 4 | 2
Not completed — Lost to Follow-up | 0 | 4 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All but one of the subjects that completed the study were included in the baseline analysis. No data was recorded for one subject who withdrew from the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Salsalate | Carvedilol | Placebo | Total
Number analyzed (Participants) | 11 | 12 | 12 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (11) | 41 (11) | 37.5 (8) | 37.5 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 2 | 15
  Male | 4 | 6 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure.
Description: Systolic blood pressure is the amount of pressure the heart generates when pumping blood through the arteries to the body. Current guidelines identify normal systolic blood pressure as lower than 120 mmHg. Blood pressure was measured in triplicate with a manual cuff prior to and every 4 hours during the 24-hour infusion with subjects in supine position. Change is the difference in systolic blood pressure at the baseline visit from pre-dosing with Intralipid to 4 hours during Intralipid infusion.
Time Frame: Pre-dose (Baseline), within 4 hours at Baseline visit
Population: One subject in the salsalate arm withdrew from the study was not included in the baseline analysis population.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 11 | 12 | 12
mmHg | 15.37 (9.15) | 10.04 (8.72) | 10.25 (12.83)

2. Primary Outcome: Change in Systolic Blood Pressure
Description: Systolic blood pressure is the amount of pressure the heart generates when pumping blood through the arteries to the body. Current guidelines identify normal systolic blood pressure as lower than 120 mmHg. Blood pressure was measured in triplicate with a manual cuff prior to and every 4 hours during the 24-hour infusion with subjects in supine position. from Change is the difference in systolic blood pressure at the baseline visit from pre-dosing with Intralipid to 8 hours during Intralipid.
Time Frame: Pre-dose (Baseline), within 8 hours at Baseline visit
Population: One subject in the salsalate arm withdrew from the study was not included in the baseline analysis population.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 11 | 12 | 12
mmHg | 13.02 (16.42) | 2.03 (11.27) | 5.47 (16.81)

3. Primary Outcome: Change in Systolic Blood Pressure
Description: Systolic blood pressure is the amount of pressure the heart generates when pumping blood through the arteries to the body. Current guidelines identify normal systolic blood pressure as lower than 120 mmHg. Blood pressure was measured in triplicate with a manual cuff prior to and every 4 hours during the 24-hour infusion with subjects in supine position. Change is the difference in systolic blood pressure at the baseline visit from pre-dosing with Intralipid to 12 hours during Intralipid infusion.
Time Frame: Pre-dose (Baseline), within 12 hours at Baseline visit
Population: One subject in the salsalate arm withdrew from the study was not included in the baseline analysis population.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 11 | 12 | 12
mmHg | 20.55 (10.06) | 1.74 (10.59) | 5.25 (15.64)

4. Primary Outcome: Change in Systolic Blood Pressure
Description: Systolic blood pressure is the amount of pressure the heart generates when pumping blood through the arteries to the body. Current guidelines identify normal systolic blood pressure as lower than 120 mmHg. Blood pressure was measured in triplicate with a manual cuff prior to and every 4 hours during the 24-hour infusion with subjects in supine position. Change is the difference in systolic blood pressure at the baseline visit from pre-dosing with Intralipid to 16 hours during Intralipid infusion.
Time Frame: Pre-dose (Baseline), within 16 hours at Baseline visit
Population: One subject in the salsalate arm withdrew from the study was not included in the baseline analysis population.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 11 | 12 | 12
mmHg | 15.78 (13.12) | 8.05 (9.35) | 3.6 (13.34)

5. Primary Outcome: Change in Systolic Blood Pressure
Description: Systolic blood pressure is the amount of pressure the heart generates when pumping blood through the arteries to the body. Current guidelines identify normal systolic blood pressure as lower than 120 mmHg. Blood pressure was measured in triplicate with a manual cuff prior to and every 4 hours during the 24-hour infusion with subjects in supine position. Change is the difference in systolic blood pressure at the baseline visit from pre-dosing with Intralipid to 20 hours during Intralipid infusion.
Time Frame: Pre-dose (Baseline), within 20 hours at Baseline visit
Population: One subject in the salsalate arm withdrew from the study was not included in the baseline analysis population.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 11 | 12 | 12
mmHg | 13.27 (9.84) | 9.39 (8.36) | 11.4 (12.70)

6. Primary Outcome: Change in Systolic Blood Pressure
Description: Systolic blood pressure is the amount of pressure the heart generates when pumping blood through the arteries to the body. Current guidelines identify normal systolic blood pressure as lower than 120 mmHg. Blood pressure was measured in triplicate with a manual cuff prior to and every 4 hours during the 24-hour infusion with subjects in supine position. Change is the difference in systolic blood pressure at the baseline visit from pre-dosing with Intralipid to 24 hours during Intralipid infusion.
Time Frame: Pre-dose (Baseline), within 24 hours at Baseline visit
Population: One subject in the salsalate arm withdrew from the study was not included in the baseline analysis population.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 11 | 12 | 12
mmHg | 13.93 (13.90) | 13.21 (11.64) | 10.27 (9.38)

7. Primary Outcome: Change in Systolic Blood Pressure
Description: Systolic blood pressure is the amount of pressure the heart generates when pumping blood through the arteries to the body. Current guidelines identify normal systolic blood pressure as lower than 120 mmHg. Blood pressure was measured in triplicate with a manual cuff prior to and every 4 hours during the 24-hour infusion with subjects in supine position. Change is the difference in systolic blood pressure at Week 6 from pre-dosing with Intralipid to 4 hours during Intralipid infusion.
Time Frame: Pre-dose (Week 6), within 4 hours at Week 6 visit
Population: 7 subjects withdrew from the study prior to the Week 6 visit. Data was also not collected for one additional subject.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 11 | 8 | 9
mmHg | 11.50 (10.54) | 14.32 (8.92) | 4.26 (13.99)

8. Primary Outcome: Change in Systolic Blood Pressure
Description: Systolic blood pressure is the amount of pressure the heart generates when pumping blood through the arteries to the body. Current guidelines identify normal systolic blood pressure as lower than 120 mmHg. Blood pressure was measured in triplicate with a manual cuff prior to and every 4 hours during the 24-hour infusion with subjects in supine position. Change is the difference in systolic blood pressure from at Week 6 from pre-dosing with Intralipid to 8 hours during Intralipid infusion.
Time Frame: Pre-dose (Week 6), within 8 hours at Week 6 visit
Population: 7 subjects withdrew from the study prior to the Week 6 visit. Data was also not collected for one additional subject.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 11 | 8 | 9
mmHg | 10.1 (11.62) | 11.62 (16.15) | 4.14 (10.43)

9. Primary Outcome: Change in Systolic Blood Pressure
Description: Systolic blood pressure is the amount of pressure the heart generates when pumping blood through the arteries to the body. Current guidelines identify normal systolic blood pressure as lower than 120 mmHg. Blood pressure was measured in triplicate with a manual cuff prior to and every 4 hours during the 24-hour infusion with subjects in supine position. Change is the difference in systolic blood pressure at Week 6 from pre-dosing with Intralipid to 12 hours during Intralipid infusion.
Time Frame: Pre-dose (Week 6), within 12 hours at Week 6 visit
Population: 7 subjects withdrew from the study prior to the Week 6 visit. Data was also not collected for one additional subject.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 11 | 8 | 9
mmHg | 9.50 (13.46) | 8.14 (15.34) | 0.38 (14.13)

10. Primary Outcome: Change in Systolic Blood Pressure
Description: Systolic blood pressure is the amount of pressure the heart generates when pumping blood through the arteries to the body. Current guidelines identify normal systolic blood pressure as lower than 120 mmHg. Blood pressure was measured in triplicate with a manual cuff prior to and every 4 hours during the 24-hour infusion with subjects in supine position. Change is the difference in systolic blood pressure at Week 6 from pre-dosing with Intralipid to 16 hours during Intralipid infusion.
Time Frame: Pre-dose (Week 6), within 16 hours at Week 6 visit
Population: 7 subjects withdrew from the study prior to the Week 6 visit. Data was also not collected for one additional subject.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 11 | 8 | 9
mmHg | 7.85 (12.60) | 7.55 (8.78) | -0.04 (6.69)

11. Primary Outcome: Change in Systolic Blood Pressure
Description: Systolic blood pressure is the amount of pressure the heart generates when pumping blood through the arteries to the body. Current guidelines identify normal systolic blood pressure as lower than 120 mmHg. Blood pressure was measured in triplicate with a manual cuff prior to and every 4 hours during the 24-hour infusion with subjects in supine position. Change is the difference in systolic blood pressure at Week 6 from pre-dosing with Intralipid to 20 hours during Intralipid infusion.
Time Frame: Pre-dose (Week 6), within 20 hours at Week 6 visit
Population: 7 subjects withdrew from the study prior to the Week 6 visit. Data was also not collected for one additional subject.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 11 | 8 | 9
mmHg | 12.88 (12.84) | 8.84 (12.25) | 6.6 (9.28)

12. Primary Outcome: Change in Systolic Blood Pressure
Description: Systolic blood pressure is the amount of pressure the heart generates when pumping blood through the arteries to the body. Current guidelines identify normal systolic blood pressure as lower than 120 mmHg. Blood pressure was measured in triplicate with a manual cuff prior to and every 4 hours during the 24-hour infusion with subjects in supine position. Change is the difference in systolic blood pressure at Week 6 from pre-dosing with Intralipid to 24 hours during Intralipid infusion.
Time Frame: Pre-dose (Week 6), within 24 hours at Week 6 visit
Population: 7 subjects withdrew from the study prior to the Week 6 visit. Data was also not collected for one additional subject.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 11 | 8 | 9
mmHg | 11.23 (9.56) | 9.92 (7.42) | 3.04 (9.41)

13. Primary Outcome: Change in Flow-mediated Dilation
Description: The change in endothelium-dependent vascular reactivity will be measured by flow-mediated dilation (FMD) of the brachial artery using a high-resolution vascular ultrasound with a 10-MHz linear array transducer. FMD is expressed as the percentage increase in diameter at the baseline visit from pre-dosing with Intralipid to 12 hours during Intralipid infusion.
Time Frame: Pre-dose (Baseline), within 12 hours at Baseline visit
Population: One subject in the salsalate arm withdrew from the study was not included in the baseline analysis population.
Measure: Mean (Standard Deviation); unit: percent change in diameter
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 11 | 12 | 12
percent change in diameter | 0.14 (0.27) | 0.24 (0.22) | 0.26 (0.34)

14. Primary Outcome: Change in Flow-mediated Dilation
Description: The change in endothelium-dependent vascular reactivity will be measured by flow-mediated dilation (FMD) of the brachial artery using a high-resolution vascular ultrasound with a 10-MHz linear array transducer. FMD is expressed as the percentage increase in diameter at the baseline visit from pre-dosing with Intralipid to 24 hours during Intralipid infusion
Time Frame: Pre-dose (Baseline), within 24 hours at Baseline visit
Population: One subject on the salsalate arm withdrew from the study was not included in the baseline analysis population.
Measure: Mean (Standard Deviation); unit: percent change in diameter
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 11 | 12 | 12
percent change in diameter | 0.35 (0.29) | 0.53 (0.47) | 0.47 (0.45)

15. Primary Outcome: Change in Flow-mediated Dilation
Description: The change in endothelium-dependent vascular reactivity will be measured by flow-mediated dilation (FMD) of the brachial artery using a high-resolution vascular ultrasound with a 10-MHz linear array transducer. FMD is expressed as the percentage increase in diameter at the Week 6 visit from pre-dosing with Intralipid to 12 hours during Intralipid infusion.
Time Frame: Pre-dose (Week 6), within 12 hours at Week 6 visit
Population: 7 subjects withdrew from the study prior to the Week 6 visit. Data was also not collected for one additional subject.
Measure: Mean (Standard Deviation); unit: percent change in diameter
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 11 | 7 | 10
percent change in diameter | 0.22 (0.27) | 0.42 (0.43) | 0.20 (0.26)

16. Primary Outcome: Change in Flow-mediated Dilation
Description: The change in endothelium-dependent vascular reactivity will be measured by flow-mediated dilation (FMD) of the brachial artery using a high-resolution vascular ultrasound with a 10-MHz linear array transducer. FMD is expressed as the percentage increase in diameter at the Week 6 visit from pre-dosing with Intralipid to 24 hours during Intralipid infusion
Time Frame: Pre-dose (Week 6), within 24 hours at Week 6 visit
Population: 7 subjects withdrew from the study prior to the Week 6 visit. Data was also not collected for one additional subject.
Measure: Mean (Standard Deviation); unit: percent change in diameter
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 11 | 7 | 10
percent change in diameter | 0.39 (0.28) | 0.70 (0.52) | 0.48 (0.29)

17. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline to 6 Weeks
Description: Diastolic blood pressure is the amount of pressure in the arteries when the heart is at rest between beats. Current guidelines identify normal diastolic blood pressure as lower than 80 mmHg. Blood pressure was measured in triplicate with a manual cuff prior to and every 4 hours during the 8 hour infusion with subjects in supine position. Change is the difference between 6-week diastolic blood pressure from baseline diastolic blood pressure.
Time Frame: Baseline, 6 weeks
Population: 6 subjects were lost to follow up, 1 withdrew from the study, and data was not collected for 1 additional subject
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 11 | 8 | 9
mmHg | 1.00 (10.13) | -1.50 (6.93) | 2.22 (10.49)

18. Secondary Outcome: Change in Oxidative Stress Markers.
Description: Oxidative stress was measured by using liquid chromatography to collect plasma glutathione and glutathione disulfide. Change is the difference between 6-week plasma glutathione and glutathione disulfide from baseline plasma glutathione and glutathione disulfide.
Time Frame: Baseline, 6 weeks
Population: not assessed (limited funds available)
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Change in Augmentation Index (AIx)
Description: AIx is a surrogate measure of peripheral arterial resistance and is measured by analysis of the pulse wave at the radial artery. The AIx is calculated as the ratio of the pulse pressure at the second systolic peak to that at the first systolic peak. Change is the difference between 6-week AIx from baseline AIx.
Time Frame: Baseline, 6 weeks
Population: not assessed (limited funds available)
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: Change in Expression of Inflammatory Biomarker Interleukin-6 (IL-6)
Description: It is measured by using microsphere-based flow cytometric immunoassay. Change is the difference between 6-week level from baseline level.
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 11 | 8 | 9
pg/ml | -0.29 (0.93) | -1.84 (5.43) | -0.36 (1.24)

21. Secondary Outcome: Change in FFA (Free Fatty Acid) Levels From Baseline to 6 Weeks
Description: Blood samples were collected for measurement of free fatty acids at baseline and 6 weeks after the Intralipid 20% infusion. FFA levels were determined by colorimetric method. Current guidelines identify normal range of FFA level as less than 0.72 mmol/L. Elevated plasma levels of FFA indicate a greater rate of insulin resistance. Change is the difference between 6-week FFA levels from baseline FFA levels.
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 11 | 8 | 9
mmol/L | -0.08 (0.32) | 0.04 (0.22) | 0.03 (0.43)

22. Secondary Outcome: Change in Pulse Wave Velocity (PWV)
Description: PWV was measured between the carotid and femoral arteries using the SphygmoCor device. Pressure waveforms at the carotid and femoral arteries were acquired using EKG gating. Velocity (distance per time in milliseconds) was calculated using the foot-to-foot method and the distance between the sites was measured manually.
Time Frame: Baseline, 6 weeks
Population: not assessed (limited funds available)
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 0 | 0 | 0

23. Secondary Outcome: Change in Expression of Inflammatory Biomarker C-Reactive Protein (CRP)
Description: It is measured by using microsphere-based flow cytometric immunoassay. Change is the difference between 6-week inflammatory biomarker level from baseline level.
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Salsalate | Carvedilol | Placebo
Number analyzed (Participants) | 11 | 8 | 9
mg/dL | 2.55 (7.67) | -7.08 (17.94) | -0.20 (2.82)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Salsalate | Carvedilol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes